CLINICAL TRIAL: NCT04695262
Title: EUS-Elastography and Contrast-Enhanced EUS Diagnostic Accuracy in the Differential Diagnosis of Subepithelial Gastrointestinal Tumors: a Multicenter Prospective Observational Study
Brief Title: EUS-Elastography and Contrast-Enhanced EUS Diagnostic Accuracy in the Differential Diagnosis of Subepithelial Gastrointestinal Tumors
Acronym: SUNNYDAY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1800
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Gastrointestinal Subepithelial Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: EUS-FNB — Endoscopic ultrasound (EUS)-guided fine needle biopsy (FNB)

SUMMARY:
The differentiation among the Gastrointestinal Subepithelial Tumors (SETs) represents a clinical challenge. Endoscopic Ultrasound (EUS) alone may be ineffective in differentiating SETs subtypes, and tissue sampling of these lesions may be technically difficult. EUS Elastography (EUS-E) has been applied to many gastrointestinal diseases, providing a qualitative/semi-quantitative stiffness analysis, but only few studies have examined the role of EUS-E in the diagnosis of SETs. In addition, the use of contrast agents has improved the diagnostic performance of the EUS, especially in the differentiation between GISTs and other gastrointestinal SETs.

The aim of the study is to examine the performance of EUS-E and Contrast Enhanced-EUS (CE-EUS) in distinguishing among different gastrointestinal SETs subtypes. EUS patterns of different techniques will be compared to the final diagnosis gained by the analysis of histopatological specimens (surgical resection or EUS-FNB) or imaging/clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GI SETs scheduled for EUS-FNB
* Patients with age > 18 but <85 years

Exclusion Criteria:

* Patients with GI SETs <15mm
* severe coagulopathy defined as abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma
* severe cardiopulmonary diseases and severe chronic kidney disease defined as glomerular filtration rate (GFR) < 15 ml/min
* known allergic disposition to SonoVue®
* pregnancy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with subepithelial gastrointestinal tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
EUS-E accuracy in terms of qualitative and quantitative elastography | 24 months
  Evaluation of EUS-E accuracy (qualitative and quantitative elastography) and contrast enhanced endoscopic ultrasound (CE-EUS) in the diagnosis of SETs.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No